CLINICAL TRIAL: NCT02817347
Title: A Randomized, Double-blind, Multicenter, Phase2 Trial to Evaluate the Safety and Efficacy of YH1177 or YH1177-D Otic Soultion in Patients With Otitis Media and Otorrhea
Brief Title: A Clinical Trial of YH1177 in Patients With Otitis Media and Otorrhea
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision for the Drug Development.
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YH1177-201
Record Dates: First submitted 2016-06-13; First posted 2016-06-29 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Otitis Media; Otorrhea
MeSH Terms: conditions — Otitis Media | interventions — Piperacillin; Tazobactam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- YH1177 (4/0.5%+0.1%) (Experimental): piperacillin 4% + tazobactam 0.5% + dexamethasone 0.1%
  Interventions: Drug: piperacillin 4% + tazobactam 0.5% + dexamethasone 0.1%
- YH1177 (8/1.0%+0.1%) (Experimental): piperacillin 8% + tazobactam 1.0% + dexamethasone 0.1%
  Interventions: Drug: piperacillin 8% + tazobactam 1.0% + dexamethasone 0.1%
- YH1177-D (2/0.25%) (Experimental): piperacillin 2% + tazobactam 0.25%
  Interventions: Drug: piperacillin 2% + tazobactam 0.25%
- YH1177-D (4/0.5%) (Experimental): piperacillin 4% + tazobactam 0.5%
  Interventions: Drug: piperacillin 4% + tazobactam 0.5%
- YH1177-D (8/1.0%) (Experimental): piperacillin 8% + tazobactam 1.0%
  Interventions: Drug: piperacillin 8% + tazobactam 1.0%

INTERVENTIONS:
Drug: piperacillin 4% + tazobactam 0.5% + dexamethasone 0.1%
  Other Names: YH1177 (4/0.5%+0.1%)
  Arms: YH1177 (4/0.5%+0.1%)
Drug: piperacillin 8% + tazobactam 1.0% + dexamethasone 0.1%
  Other Names: YH1177 (8/1.0%+0.1%)
  Arms: YH1177 (8/1.0%+0.1%)
Drug: piperacillin 2% + tazobactam 0.25%
  Other Names: YH1177-D (2/0.25%)
  Arms: YH1177-D (2/0.25%)
Drug: piperacillin 4% + tazobactam 0.5%
  Other Names: YH1177-D (4/0.5%)
  Arms: YH1177-D (4/0.5%)
Drug: piperacillin 8% + tazobactam 1.0%
  Other Names: YH1177-D (8/1.0 %)
  Arms: YH1177-D (8/1.0%)

SUMMARY:
In patients with otitis media presenting with otoscopy-confirmed otorrhea who had tympanostomy tube insertion or tympanic perforation, to evaluate the safety, tolerability, and the proportion of patients with cessation of otorrhea after ear-drop administration of YH1177 or YH1177-D for 14 days and therefore to determine the optimal clinical dose.

DETAILED DESCRIPTION:
Patients with otitis media presenting with otoscopy-confirmed otorrhea who had tympanostomy tube insertion or tympanic perforation. Screening should be completed within 7 days prior to randomization.

patients with otitis media presenting with otoscopy-confirmed otorrhea who had tympanostomy tube insertion or tympanic perforation at randomization visit will be randomized in one of the defined groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent A detailed explanation about the study, including the study purpose and procedures and drug properties, had been provided, and the patient gave voluntary written informed consent.
* Target Population Patients with otitis media presenting with otorrhea, as evidenced by otoscopy, who had tympanostomy tube insertion or tympanic perforation
* Sex and age Male or female patients 19 years of age or older at screening Women of childbearing potential (WOCBP) must have 'negative' pregnancy test at screening, and use an acceptable method of contraception throughout the study.

Exclusion Criteria:

* Excluded Disease

  1. Patients diagnosed with otitis media with cholesteatoma, otitis media with effusion or otitis externa at screening
  2. Patients who had a otologic surgery within 1 year prior to screening (except for tympanostomy tube insertion)
  3. Subjects who previously had cholesteatoma or mastoid surgery
* Medical History and Concurrent Disease

  1. Patients with complication of labyrinthine fistula at screening
  2. Patients with clinically significant medical or mental illness.
  3. Patients with infectious disease requiring the use of systemic antimicrobial therapy
* Physical and Laboratory Test Results

  a)Clinically significant finding based on the principal investigator/investigator's opinion.
* Allergies and Adverse Drug Reactions

  1. Known drug allergy (e.g., a history of anaphylaxis or hepatotoxicity)
  2. History of hypersensitivity to penicillins or -lactamase inhibitors.
  3. History of serious skin reaction such as Stevens-Johnson syndrome or toxic epidermal necrosis
* Prohibited Therapies and/or Medication

  1. Patients undergoing a ventilation tube insertion on the day of screening
  2. Patients with ventilation tube containing silver oxide or silver salt (e.g., T-type tube)
* Reproductive status, Women only

  a)Woman of childbearing potential (WOCBP) who is unable, or unwilling to use an acceptable method of contraception during the study
* Other Exclusion Criteria

  1. History of alcohol or drug abuse/addiction within the last 1 year prior to the study entry
  2. Patient who, in the investigator's opinion, is not suitable for the study for any reason (e.g., ECG or hepatitis test results at screening)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving cessation of otorrhea on Day 15. | Day 15
  The proportion of patients achieving cessation of otorrhea (grade 0) on Day 15, as evidenced by otoscopy

SECONDARY OUTCOMES:
The proportion of patients with cessation of otorrhea on Day 8. | Day 8
  The proportion of patients with cessation of otorrhea on Day 8 as evidenced by otoscopy.
The proportion of patients with cessation of otorrhea on Day 22. | Day 22
  The proportion of patients with cessation of otorrhea on Day 22 as evidenced by otoscopy.
Proportion of patients with improved otorrhea at each visit, as evidenced by otoscopy | Day 8
  'improved otorrhea' is defined as at least one level decrease from baseline in the otorrhea severity grading scale
Proportion of patients with improved otorrhea at each visit, as evidenced by otoscopy | Day 15
  'improved otorrhea' is defined as at least one level decrease from baseline in the otorrhea severity grading scale
Proportion of patients with improved otorrhea at each visit, as evidenced by otoscopy | Day 22
  'improved otorrhea' is defined as at least one level decrease from baseline in the otorrhea severity grading scale
Microbiological eradication | Day 8, 15, 22
  Proportion of patients with microbiological eradicationat each visit

OTHER OUTCOMES:
Cmax | pre-dose, and at 0.25, 0.5, 1, 2, 4 and 6 hours
  Maximum plasma concentration
AUClast | pre-dose, and at 0.25, 0.5, 1, 2, 4 and 6 hours
  The area under the plasma concentration-time curve from time zero until the last measurable concentration
AUCinf | pre-dose, and at 0.25, 0.5, 1, 2, 4 and 6 hours
  The area under the plasma concentration - time curve from time zero to infinite time
Tmax | pre-dose, and at 0.25, 0.5, 1, 2, 4 and 6 hours
  Time to reach Cmax
t1/2 | pre-dose, and at 0.25, 0.5, 1, 2, 4 and 6 hours
  Terminal elimination half-life
CL/F | pre-dose, and at 0.25, 0.5, 1, 2, 4 and 6 hours
  Apparent plasma clearance
Vd/F | pre-dose, and at 0.25, 0.5, 1, 2, 4 and 6 hours
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: chulho jang, M.D Ph.D, Study Chair — Chonnam National Universitiy Hospital
Locations (1):
- Chonnam National Universitiy Hospital, Gwangju, Chonnam, South Korea